CLINICAL TRIAL: NCT02316418
Title: Prospective Safety and Efficacy Evaluation of Hairstetics™ Anchoring System for Hair Extensions in Female Pattern Hair Loss
Brief Title: Hairstetics™ Anchoring System in Female Pattern Hair Loss (HAS-FPHL)
Acronym: HAS-FPHL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hairstetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HET-11
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Female Pattern Baldness; Alopecia, Androgenetic
Keywords: Hairstetics™ anchoring system; hair extensions
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hairstetics™ anchoring system (Experimental): Prosthetic hair implantation using the Hairstetics™ anchoring system, followed by attachment of hair extensions.
  Interventions: Device: Hairstetics™ anchoring system

INTERVENTIONS:
Device: Hairstetics™ anchoring system — Overall, up to 360 prosthetic hair implants will be set in the scalp. The procedure will be performed in accordance with the instructions in the device Instructions for Use. Training and certification of operators by the Sponsor is a prerequisite for use of the study device by the former.
  Hair extensions will be attached to the fibers four weeks after the implantation.

SUMMARY:
The aim of the study is to provide evidence of safety and preliminary performance of the Hairstetics™ anchoring system in female subjects affected with androgenetic alopecia (female pattern hair loss; (FPHL)).

The study will also help to determine whether the Hairstetics™ anchoring system, in conjunction with attachment of hair extensions, is efficacious in improving patient and physician aesthetic satisfaction with the treated scalp appearance in female patients with androgenetic alopecia.

DETAILED DESCRIPTION:
* Type of trial: Open label
* Study population: Female patients with androgenetic alopecia (FPHL)
* Phase: II
* Number of study arms: Single-arm
* Number of centers: Single center
* Name of study agent: Hairstetics™ hair anchoring system
* Changes in scheduling: maximal number of implants may not be modified throughout the trial.

ENDPOINTS

Primary Endpoint:

Percent of subjects with at least 70% of the hair extensions remaining in place at the 6-month follow-up visit.

Secondary Endpoints:

* Proportion of hair extensions remaining at place at the different visits.
* Subject aesthetic satisfaction based on a satisfaction questionnaire (on a scale of 1-10).
* Investigator aesthetic satisfaction based on a satisfaction questionnaire on a scale of 1-10).
* Pain rating during procedure, based on a visual analogue numeric pain rating scale (on a scale of 0-10).

Exploratory Endpoints:

* Ease of use, based on a user questionnaire responses (on a scale of 1-10).
* Implant retrieval rate.

Safety Endpoints:

Adverse events both expected and unexpected, related or unrelated to study device or procedure, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03.

STUDY PROCEDURE - After signing informed consent, patients will be screened for study eligibility by assessment of inclusion and exclusion criteria. Screening procedures will include collection of demographic data, medical history, physical examination, vital signs, and laboratory evaluations.

Unless the patient's participation in the trial is terminated, subjects will then be implanted with Hairstetics™ anchoring system cartridges holding up to a total of 360 of the Hairstetics™ prosthetic hair units. Complete blood count (CBC), biochemistry and coagulation panel and a quantitative β-HCG, as specified in the eligibility criteria, will be required before treatment and the test requirements specified in the inclusion criteria must be met.

Patients will be followed a week after the study implantation procedure, to ensure proper monitoring of safety events.

Hair extensions will be attached four weeks after the implantation. Patients will be followed at 3 and 6 months after the attachment of hair extensions.

This protocol will allow excision of implants.

This protocol does not provide arrangements for long-term follow-up of study participants beyond primary endpoint.

SUBJECT POPULATION - Female patients with androgenetic alopecia (female pattern hair loss; (FPHL))

STUDY DURATION - 13 months.

STATISTICAL ANALYSIS - General -

No separate Statistical Analysis Plan (SAP) document is planned. Nevertheless, if during the study, modifications to the statistical considerations will be deemed necessary, a SAP may be issued.

The study is planned as a prospective, single-arm study to assess safety and preliminary efficacy data on the treatment of female subjects affected with androgenetic alopecia (FPHL) with the Hairstetics™ anchoring system. The analysis of the endpoints is descriptive in nature; no formal statistical hypotheses will be tested.

Primary Endpoint:

The number and proportion of subjects with at least 70% of the hair extensions remaining in place at the 6-month follow-up visit, will be presented.

Secondary Endpoints:

The proportion of hair extensions remaining in place at the different visit will be presented in a tabular form.

The aesthetic satisfaction as assessed by the subjects and the investigators will be presented in a tabular form by visit, once as continuous variables, and once as categorical variables.

The pain during the procedure will be presented in a tabular form, once as continuous variable, and once as categorical variable.

Exploratory analyses:

The ease of use will be presented in the same manner as the pain. The number and proportion of subjects for whom the implants are removed will be presented in a tabular form.

Safety endpoint:

The cumulative incidence (and 95% CI) of adverse events observed during procedure and throughout the follow-up period, will be presented in tabular format. A detailed list of all adverse events will be presented. The adverse event rate will be compiled with respect to seriousness, severity, and relationship to procedure and device. In addition, listings of all safety measures will be produced.

Baseline descriptive statistics:

Demographic, medical and clinical history variables will be tabulated. Continuous variables will be summarized by a mean, standard deviation, minimum, median and maximum, and categorical variables by a count and percentage.

Interim analysis:

No interim analysis is planned for efficacy and/or safety review.

Sample size:

No formal sample size calculations were performed. A sample size of ten subjects will provide safety and performance preliminary assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 yrs.
2. Female patients with androgenetic alopecia (FPHL).
3. Pre-treatment hematology and coagulation values within the limits:

   1. Hemoglobin ≥ 10 g/dl (g/100 ml)
   2. Platelets ≥ 150 x 10^9/L (10^3/mm^3)
   3. WBC ≥ 3.0 x 10^9/L (10^3/mm^3)
   4. INR 0.8 - 1.2 ---
   5. PTT 25" - 35"
   6. Serum creatinine < 2 mg/dl
   7. SGOT < 1.5 x ULN (Upper Limit of Norm)
   8. SGPT < 1.5 x ULN
   9. Alkaline phosphatase < 1.5 x ULN
4. A life expectancy at least of the duration of the trial.
5. Signed informed consent and post-implantation protocol.

Exclusion Criteria:

1. Prosthetic hair implantation or hair transplantation in the 6 months preceding enrollment to this study.
2. Skin conditions that might affect the procedure and/or its outcome. NOTE: Such conditions are not necessarily restricted to or involve the prospective implantation site and/or its vicinity.
3. Patients currently receiving, or that have received within the past 3 months, radio- and/or chemotherapy.
4. Patients on anticoagulant treatment.
5. More than a maintenance dose of oral corticosteroids (maintenance dose is defined as the same dose regimen over the past 6 months for a condition requiring continual corticosteroid treatment) or patients with an immunocompromised state for any reason.
6. Bleeding disorder.
7. Patient presenting with a health condition that may affect compliance with the study protocol, either by itself or combined with other conditions present in the patient.
8. Use of illegal substances.
9. Participation in another interventional study, unless discussed with and approved by the Sponsor or Sponsor's authorized representative.
10. Quantitative β-HCG ≥ 5 mIU/mL (IU/L) in women of childbearing potential.
11. Lactating and/or breastfeeding women.
12. Known hypersensitivity (e.g., to nitinol, nickel or titanium) or adverse event that would prevent a prospective study participant from being administered the trial treatment or non-investigational medicinal product(s), as detailed in the protocol.
13. Patients with implanted electronic devices (such as cardiac pacemakers) unless they receive permission from their treating physician (e.g., cardiologist) and are monitored by a treating physician during the treatment session.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-02 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects with at least 70% of the hair extensions | 6 months after attachment of hair extensions
  Percent of subjects with at least 70% of the hair extensions remaining in place at the 6-month follow-up visit.

SECONDARY OUTCOMES:
Subject aesthetic satisfaction | at the time of enrolment, after attaching hair extensions and 3 and 6 months after the study treatment
  Satisfaction of study participants with the aesthetic appearance of their scalp will be assessed through a questionnaire. Participants will provide a numerical evaluation, on a standard scale of 1-10, of their satisfaction (with 10 being the highest grade of satisfaction).
Investigator aesthetic satisfaction | at the time of enrolment, after attaching hair extensions and 3 and 6 months after the study treatment
  Satisfaction of Investigators with the aesthetic appearance of the scalp of study subjects will be assessed. Investigators will provide a numerical evaluation, on a standard scale of 1-10, of their satisfaction (with 10 being the highest grade of satisfaction). Digital photography and, optionally, video will be used throughout the study, starting with the screening and during every visit thereafter, to capture the general appearance of the scalp and that of the implantation area and its vicinity. Digital images may support Investigators in providing their evaluation of the procedural outcome.
Proportion of hair extensions remaining at place at the different visits. | from attachment of hair extensions through study completion, an average of 6 months
Pain rating during procedure | At implantation
  Pain rating, based on a visual analogue numeric pain rating scale (on a scale of 0-10).

OTHER OUTCOMES:
Device ease of use | At implantation
  Ease of use of the device, based on a user questionnaire responses (on a scale of 1-10).
Implant retrieval rate | from implantation through study completion, an average of 7 months
Cumulative incidence of adverse events | through study completion, an average of 7.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Igal Ruvinsky, Ph.D., Study Director — Hairstetics Ltd.
Locations (1):
- Fortis Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No